CLINICAL TRIAL: NCT07177443
Title: Induction Chemotherapy Combined With Serplulimab Induction/Maintenance Therapy and Omission of Concurrent Chemotherapy in Locally Advanced Nasopharyngeal Carcinoma (UNION-NPC-001): A Multicenter, Open-Label, Randomized, Controlled, Phase III, Non-Inferiority Clinical Trial
Brief Title: Serplulimab Combined With Induction Chemotherapy and Radiotherapy in Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNION-NPC-001
Record Dates: First submitted 2025-08-05; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
Keywords: Cisplatin-based concurrent chemoradiotherapy; radiotherapy; Treatment De-escalation; locally advanced nasopharyngeal carcinoma
MeSH Terms: interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Radiotherapy
  Interventions: Radiation: Radiotherapy; Drug: Serplulimab
- Control arm (Active Comparator): Cisplatin-based concurrent chemoradiotherapy (CCRT)
  Interventions: Radiation: Radiotherapy; Drug: Serplulimab; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiotherapy — Following induction therapy, eligible patients will receive radiotherapy alone or concurrent chemoradiotherapy per protocol. Photon or proton radiotherapy techniques were permitted. Prescribed doses were:
  Primary tumor and metastatic lymph nodes: 70 Gy/33 fractions High-risk lymphatic drainage areas: 60 Gy/33 fractions Low-risk regions: 54 Gy/33 fractions
  PTV dose specifications:
  GTVnx: 70 Gy GTVnd: 66-70 Gy (reducible to 63 Gy for suspicious small nodes) CTV1: 60-62 Gy CTV2: 54-56 Gy All treatments will employ simultaneous integrated boost (SIB) intensity-modulated radiotherapy delivered once daily, 5 fractions per week.
Drug: Serplulimab — Serplulimab will be used in the induction phase for 3 cycles and the maintenance phase for 14 cycles.
Drug: Cisplatin — On days 64 and 85, patients will receive cisplatin chemotherapy at a dose of 100 mg/m² via intravenous infusion.
  Arms: Control arm

SUMMARY:
This phase III trial aims to evaluate the efficacy and safety of induction chemotherapy combined with serplulimab (induction/maintenance therapy) with omission of concurrent chemotherapy in patients with locally advanced nasopharyngeal carcinoma (LA-NPC).

DETAILED DESCRIPTION:
This multicenter phase III trial enrolls high-risk locally advanced nasopharyngeal carcinoma patients (AJCC 9th edition, Stage T1-3N2 [II] or T1-4N3/T4N1-2 [III]) who achieves ≥50% tumor regression (RECIST v1.1) and undetectable plasma EBV DNA after three cycles of GP induction chemotherapy (gemcitabine + cisplatin) combined with serplulimab. Eligible patients will be randomized to either:

Experimental arm: Radiotherapy alone followed by serplulimab maintenance, or Control arm: Cisplatin-based concurrent chemoradiotherapy (CCRT) followed by serplulimab maintenance.

Primary study endpoint

* 3-year event-free survival (EFS)

  * 5-year overall survival (OS)

    * incidence of treatment-induced vomiting Secondary study endpoints
* 3-year distant metastasis-free survival (DMFS)

  * 3-year locoregional recurrence-free survival (LRFS)

    * Quality of life (QoL) assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30 v3.0) and its head-and-neck cancer module (EORTC QLQ-H&N35 v1.0), both validated Chinese versions.

      * Incidence rate of investigator-reported adverse events (AEs) ⑤ Incidence rate of patient-reported AEs

ELIGIBILITY:
Inclusion Criteria:

1. Age at diagnosis: 18-65 years;
2. Pathologically confirmed treatment-naïve nasopharyngeal carcinoma of "non-keratinizing type (WHO classification)";
3. Locoregionally advanced nasopharyngeal carcinoma staged per the 9th edition of the American Joint Committee on Cancer (AJCC) staging system: Stage II (T1-3N2), Stage III(T1-4N3 or T4N1-2);
4. ECOG performance status: 0-1;
5. Post-induction therapy requirements:

   Radiological assessment showing ≥50% tumor regression (RECIST 1.1) Undetectable plasma EBV DNA levels;
6. Adequate bone marrow function:

   White blood cell count >4×10⁹/L Hemoglobin >90 g/L Platelet count >100×10⁹/L;
7. Normal hepatic/renal function:

   Total bilirubin ≤1.5×upper limit of normal (ULN) AST/ALT ≤2.5×ULN Alkaline phosphatase ≤2.5×ULN Creatinine clearance ≥60 mL/min;
8. Normal results for:

   Thyroid function tests Amylase and lipase Pituitary function Inflammatory/infection markers Cardiac enzymes Electrocardiogram

   Additional requirements:

   Pulmonary function tests for smokers >50 years Cardiac ultrasound + myocardial function tests for patients with ECG abnormalities or cardiovascular history (unless meeting exclusion criterion (8));
9. Signed informed consent with willingness/compliance to follow study schedules for treatment, follow-up, and laboratory tests;
10. For women of childbearing potential: Agreement to use reliable contraception (e.g., condoms, prescribed oral contraceptives) from screening until 1 year post-treatment.

Exclusion Criteria:

1. Hepatitis B Virus (HBV) Infection:

   HBsAg-positive with HBV DNA >1×10³ copies/mL (patients with controlled viremia [<1×10³ copies/mL] after antiviral therapy are eligible).
2. Hepatitis C Virus (HCV) Infection: Anti-HCV antibody-positive.
3. HIV/AIDS: Anti-HIV antibody-positive or diagnosed with acquired immunodeficiency syndrome (AIDS).
4. Active Tuberculosis (TB): History of active TB within the past year (regardless of treatment status). Exception: Patients with adequately treated past TB (confirmed by standard anti-TB therapy) may be enrolled if >1 year since completion of treatment.
5. Active Autoimmune Diseases:Known or suspected autoimmune disorders (e.g., uveitis, colitis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, hypothyroidism, or asthma requiring bronchodilators).

   Exceptions:

   Type 1 diabetes mellitus Hypothyroidism managed with hormone replacement Skin conditions not requiring systemic therapy (e.g., vitiligo, psoriasis, alopecia).
6. Interstitial Lung Disease (ILD):

   History of ILD or pneumonitis requiring oral/IV steroids within the past year.
7. Immunosuppressive Therapy:

   Chronic systemic corticosteroids (≥10 mg prednisone equivalent/day) or other immunosuppressants within 4 weeks prior to enrollment. Inhaled/topical steroids are permitted.
8. Uncontrolled Cardiac Disease: Heart failure (NYHA class ≥2), Unstable angina, Myocardial infarction within the past year, Clinically significant arrhythmias requiring treatment.
9. Pregnancy/Lactation: Pregnant or breastfeeding women (urine/blood pregnancy test required for women of childbearing potential).
10. Concurrent Malignancies:

    History of other malignancies except:

    Adequately treated non-melanoma skin cancer, Carcinoma in situ of the cervix, Papillary thyroid carcinoma.
11. Hypersensitivity: Known allergy to any component of the study drugs or excipients.
12. Active Infections:

    Systemic infections requiring treatment within 1 week prior to enrollment.

    Live Vaccines:
13. Administration of live vaccines within 30 days before the first immunotherapy dose.
14. Organ Transplantation: History of allogeneic organ transplantation.
15. Other High-Risk Conditions:

Any condition that may compromise patient safety or compliance per investigator assessment (e.g., severe psychiatric disorders, life-threatening comorbidities, or social/familial risk factors).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 3-year
  EFS is defined as the time from the date of randomization to the first occurrence of disease recurrence (locoregional or distant) or death from any cause, whichever comes first.
Overall survival (OS) | 5-year
  OS is defined as the time from the date of randomization until death from any cause.
Incidence rate of all-grade vomiting | Through study completion, an average of 1 year
  Incidence rate of all-grade vomiting during treatment assessed by clinicians according to the Common Terminology Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Distant metastasis-free survival (DMFS) | 3-year
  DMFS is defined as the time from the date of randomization to the first radiological or pathological confirmation of distant metastasis.
Locoregional recurrence-free survival (LRFS) | 3-year
  LRFS is defined as the time from the date of randomization to the first histologically or radiologically confirmed locoregional recurrence.
Health-Related Quality of Life assessed by EORTC QLQ-C30 | From baseline (at informed consent) up to 60 months after radiotherapy completion.
  Changes in health-related quality of life from baseline (informed consent) until 60 months after radiotherapy completion, assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), version 3.0. The QLQ-C30 includes functional scales (e.g., physical, role, emotional), global quality of life scale, and symptom scales (e.g., fatigue, pain, nausea/vomiting). Scores range from 0 to 100. For functional scales and global quality of life, a higher score represents a better level of functioning or well-being. For symptom scales, a higher score represents a greater severity of symptoms.
Head and Neck Cancer-Specific Symptoms assessed by EORTC QLQ-H&N35 | From baseline (informed consent) until 60 months after radiotherapy completion.
  Changes in head and neck cancer-specific symptoms and side effects from baseline (informed consent) until 60 months after radiotherapy completion, assessed using the EORTC Head and Neck Cancer Module (QLQ-H&N35), version 1.0. The QLQ-H&N35 assesses symptoms relevant to head and neck cancer patients (e.g., pain, swallowing, senses, speech, social eating). Scores range from 0 to 100. For all symptom scales, a higher score represents a greater severity of symptoms.
Incidence rate of investigator-reported adverse events (AEs) | 3-year
  Analysis of investigator-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0.
Incidence rate of patient-reported adverse events (AEs) | 3-year
  Analysis of patient-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by patients themselves

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No